CLINICAL TRIAL: NCT00780949
Title: Immunological Consequences of CARD15/NOD2 Mutations in Crohn's Disease
Acronym: PLAC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: P071206
Record Dates: First submitted 2008-10-27; First posted 2008-10-28 (Estimated); Last update posted 2012-08-03 (Estimated); Status verified 2012-07

CONDITIONS: Crohn's Disease
Keywords: Crohn's Disease, inflammatory bowel disease, Peyer's patches
MeSH Terms: conditions — Crohn Disease; Inflammatory Bowel Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1: Crohn's disease patient (Experimental): intestinal biopsies
  Interventions: Other: intestinal biopsies

INTERVENTIONS:
Other: intestinal biopsies — intestinal biopsies during routine endoscopy
  Other Names: intestinal biopsies during routine endoscopy

SUMMARY:
The project is based on adult and paediatric cohorts among the largest ones in Paris and located at Saint Louis and Robert Debré hospitals. Experiments will be performed at INSERM Unit U843 in collaboration with the department of immunology and statistics, Robert Debré Hospital.

DETAILED DESCRIPTION:
Crohn's Disease (CD) affects about 60.000 to 80.000 people in France. It is characterised by a chronic or relapsing inflammation of the gut. Its aetiology is largely unknown, limiting the development of preventive and curative therapeutic options. In 2001, we have identified the first CD susceptibility gene: CARD15/NOD2. This gene is involved in the innate immune response but we do not know today how gene mutations may induce the disease lesions. However, many data suggest that the intestinal inflammation may be related with an abnormal function of the lymphoid tissue present in the gut.

The aim of the present proposal is to better understand the role of CARD15/NOD2 mutations (R702W, G908R and 1007fs) in the development and the function of the intestinal lymphoid tissue. 250 patients and controls will be enrolled at Robert Debré and Saint Louis Hospital (Paris, France) within a 2 years period.

For participant, 4 to 5 ileal biopsies will be taken during a routine colonoscopy. Patients will be classed in three groups according to their number of CARD15/NOD2 mutations (1) wild-type, 2) mutated heterozygotes and 3) mutated homozygotes or compound heterozygotes). A comparison between groups and with non inflammatory (colonoscopy performed for other reasons) or inflammatory (ulcerative colitis patients) controls will be done. For each group, cell phenotype, cytokine profile, permeability and bacterial translocation will be analysed on Peyer's patches.

The project is based on adult and paediatric cohorts among the largest ones in Paris and located at Saint Louis and Robert Debré hospitals. Experiments will be performed at INSERM Unit U843 in collaboration with the department of immunology and statistics, Robert Debré Hospital.

ELIGIBILITY:
Inclusion Criteria:

* Children and adults ≥ 5 ans and ≤ 65 ans with a programmed routine colonoscopy for Crohn's disease, ulcerative colitis, or another benign gastroenterological disorder

Exclusion Criteria:

* Patients < 5 ans or > 65 ans
* Patients with contra-indications for multiple biopsies
* Patients with an undeterminate colitis

Ages: 5 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2009-01; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
cytokine production and cell phenotype in Peyer patches | final time frame at the end of the study

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Pierre HUGOT, Professeur, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hopital Robert Debre, Paris, France